CLINICAL TRIAL: NCT01100905
Title: Utility of an Iron-containing Food Product for the Prevention of Diminished Iron Status During Basic Combat Training
Brief Title: An Iron-containing Food Product for the Prevention of Diminished Iron Status in Soldiers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: James P. McClung, Ph.D., USARIEM
Other Study IDs: H08-11
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Iron Deficiency; Iron Deficiency Anemia
Keywords: Iron; Iron status; Iron deficiency; Iron deficiency anemia
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Iron-containing food product

SUMMARY:
Military personnel face intense physical and cognitive demands. Diminished iron status affects physiologic responses to these challenges. Both cross-sectional and longitudinal studies indicate a significant decrement in iron status in enlisted female military personnel immediately following basic combat training (BCT). Decrements in iron status are associated with diminished cognitive and physical performance, and may affect body composition. The primary objective of this randomized, placebo controlled study is to assess the utility of an iron-containing food product for maintaining iron status during BCT. This study will provide insight into the utility and efficacy of an iron-containing food product for the maintenance of iron status during military training. Furthermore, it will provide novel scientific data regarding the relationship between iron status and physical and cognitive performance in female Soldiers.

ELIGIBILITY:
Inclusion Criteria:

* Female US Army Recruit
* Participating in Basic Combat Training

Exclusion Criteria:

* Male
* Pregnancy
* Diagnosed hemochromatosis
* Diagnosed thalassemia
* History of ulcerative colitis
* Allergy to chocolate

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Fort Jackson, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Karl JP, Lieberman HR, Cable SJ, Williams KW, Young AJ, McClung JP. Randomized, double-blind, placebo-controlled trial of an iron-fortified food product in female soldiers during military training: relations between iron status, serum hepcidin, and inflammation. Am J Clin Nutr. 2010 Jul;92(1):93-100. doi: 10.3945/ajcn.2010.29185. Epub 2010 May 5. PMID 20444958